CLINICAL TRIAL: NCT04195308
Title: Accelerated Intermittent Theta-burst Stimulation for Treatment of Preoperative Depression to Reduce Conversion of Acute to Chronic Opioid Use Following Arthroplasty
Brief Title: SAINT for Treatment of Preoperative Depression to Reduce Opioid Use Following Arthroplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical constraints
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Nolan R, Assistant Professor, Department of Psychiatry and Behavioral Sciences, Stanford University, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-53022
Record Dates: First submitted 2019-10-25; First posted 2019-12-11 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Treatment Resistant Depression
Keywords: transcranial magnetic stimulation; theta burst
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TBS-DLPFC (Experimental): The active group will receive theta-burst TMS stimulation.
  Interventions: Device: Active TBS-DLPFC
- Sham TBS-DLPFC (Sham Comparator): The sham group will receive sham theta-burst TMS stimulation. Participants will have the option of open label TBS-DLPFC treatment following study completion.
  Interventions: Device: Sham TBS-DLPFC; Device: Open label TBS-DLPFC

INTERVENTIONS:
Device: Active TBS-DLPFC — Participants in the active stimulation group will receive intermittent TBS to left DLPFC. The L-DLPFC will be targeted utilizing the Localite neuronavigation system. Stimulation intensity will be standardized at 90% of RMT and adjusted to the skull to cortical surface distance (see Nahas 2004).
  Stimulation will be delivered to the L-DLPFC using a MagPro stimulator.
  Arms: Active TBS-DLPFC
Device: Sham TBS-DLPFC — The parameters in the active arms will be as above with the internal randomization of the device internally switching to sham in a blinded fashion.
  Arms: Sham TBS-DLPFC
Device: Open label TBS-DLPFC — Patients will have the option of receiving active, open label aTBS treatment following sham.
  Stimulation will be delivered to the L-DLPFC using a MagPro stimulator or Nexstim TMS device.
  Arms: Sham TBS-DLPFC

SUMMARY:
This study evaluates an accelerated schedule of theta-burst stimulation using a transcranial magnetic stimulation device for treatment-resistant depression. In a double-blind fashion, half the participants will receive accelerated theta-burst stimulation while half will receive sham treatment.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is an established technology as therapy for treatment-resistant depression. The approved method for treatment is 10Hz stimulation for 40 min over the left dorsolateral prefrontal cortex (L-DLPFC). This methodology has been effective in real world situations. The limitations of this approach include the duration of the treatment (approximately 40 minutes per treatment session, 5 days per week, for 4-8 weeks). Recently, researchers have pursued modifying the treatment parameters to reduce treatment times with some preliminary successes. This study aims to further modify the parameters to create a more rapid form of the treatment and look at the change in neuroimaging biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 22 to 80 years of age.
* Able to provide informed consent.
* Diagnosed with Major Depressive Disorder (MDD) and currently experiencing a Major Depressive Episode (MDE).
* Participants may currently be on a stable and adequate dose of SSRI antidepressant therapy. Participants may choose to not be on antidepressant therapy for the study duration, or to be switched from other classes to a medication from the SSRI class.
* Participants may also have a history of intolerance to at least 2 antidepressant medications. These patients with the intolerance history will not be required to be currently taking an antidepressant medication.
* Participants must qualify as "Moderately Treatment Refractory" or "High Treatment Refractory" using the Maudsley staging method.
* Meet the threshold on the total HAMD17 score of >/=20 at both screening and baseline visits (Day -5/-14 and Day 0).
* Meet the threshold on the total MADRS score of >/=20 at both screening and baseline visits (Day -5/-14 and Day 0).
* Meet the threshold on the total BDI-II score of >/=20 at both screening and baseline visits (Day -5/-14 and Day 0).
* In good general health, as ascertained by medical history.
* If female, a status of non-childbearing potential or use of an acceptable form of birth control. The form of birth control will be documented at screening and baseline.
* Concurrent hypnotic therapy (e.g., with zolpidem, zaleplon, melatonin, or trazodone) will be allowed if the therapy has been stable for at least 4 weeks prior to screening and if it is expected to remain stable.

Exclusion Criteria:

* Female of childbearing potential who is not willing to use one of the specified forms of birth control during the study.
* Female that is pregnant or breastfeeding.
* Female with a positive pregnancy test at participation.
* Total HAMD17 score of < 20 at the screen or baseline visits.
* Total MADRS score of < 20 at the screen or baseline visits.
* Total BDI-II score of < 20 at the screen or baseline visits.
* Current diagnosis of a Substance Use Disorder (Abuse or Dependence, as defined by DSM-IV-TR), with the exception of nicotine dependence, at screening or within six months prior to screening.
* Current diagnosis of Axis I disorders other than Dysthymic Disorder, Generalized Anxiety Disorder, Social Anxiety Disorder, Panic Disorder, Agoraphobia, or Specific Phobia (unless one of these is comorbid and clinically unstable, and/or the focus of the participant's treatment for the past six months or more).
* History of schizophrenia or schizoaffective disorders, or any history of psychotic symptoms in the current or previous depressive episodes.
* Any Axis I or Axis II Disorder, which at screening is clinically predominant to their MDD or has been predominant to their MDD at any time within six months prior to screening.
* Considered at significant risk for suicide during the course of the study.
* Has a clinically significant abnormality on the screening examination that might affect safety, study participation, or confound interpretation of study results.
* Participation in any clinical trial with an investigational drug or device within the past month or concurrent to study participation.
* Any current or past history of any physical condition which in the investigator's opinion might put the subject at risk or interfere with study results interpretation.
* History of positive screening urine test for drugs of abuse at screening: cocaine, amphetamines, barbiturates, opiates.
* Current (or chronic) use of opiates.
* History of epilepsy.
* History of rTMS exposure.
* History of any implanted device or psychosurgery for depression.
* History of ECT intolerance.
* History of shrapnel or metal in the head or skull.
* "Low Treatment Refractory" using the Maudsley staging method.
* History of cardiovascular disease or cardiac event.
* History of OCD.
* History of autism spectrum disorder.
* History of intractable migraine
* History of independent sleep disorder.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery-Åsberg Depression Rating Scale (MADRS) score from pre-treatment to 1-month post-treatment. | Pretreatment to 1-month posttreatment
  A ten item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders.

SECONDARY OUTCOMES:
Percentage change in the Hamilton Rating Scale for Depression (HAMD-17) | 4 weeks posttreatment
  A provider administered questionnaire used to assess remission and recovery from depression.
Percentage change in the Columbia Suicide Severity Rating Scale (C-SSRS) | Pretreatment, immediately posttreatment, 2 weeks posttreatment, 4 weeks posttreatment
  A suicidal ideation rating scale created by researchers at Columbia University.
Percentage change in the Hamilton Rating Scale for Depression (HAM-6) | Follow-up every 2 weeks for 6 months by telephone
  A 6 item questionnaire used to score the severity of depression.
Percentage change in the Hamilton Rating Scale for Depression (HAMD-17) | Pretreatment, immediately posttreatment, 2 weeks posttreatment
  A provider administered questionnaire used to assess remission and recovery from depression.
Change in baseline functional connectivity to immediate post-treatment using functional MRI | Pretreatment to immediately posttreatment
  MR imaging of the brain to measure the functional connectivity between the subcallosal cingulate to the default mode network.
Change in baseline functional connectivity to 1-month post-treatment | Pretreatment to 1-month post-treatment
  The investigators will assess functional connectivity as seen on resting state fMRI, between the subcallosal cingulate to the default mode network and within the default mode network.
Change in baseline heart rate variability through immediate post treatment and 1-month post treatment | Pretreatment, immediately posttreatment and 1-month post treatment
  Heart rate variability measures will be compared baseline, immediate post treatment and 1-month post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nolan Williams, MD, Principal Investigator — Stanford University
Locations (1):
- Department of Psychiatry and Behavioral Sciences, Stanford School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Background] George MS, Wassermann EM, Williams WA, Callahan A, Ketter TA, Basser P, Hallett M, Post RM. Daily repetitive transcranial magnetic stimulation (rTMS) improves mood in depression. Neuroreport. 1995 Oct 2;6(14):1853-6. doi: 10.1097/00001756-199510020-00008. PMID 8547583
- [Background] Pascual-Leone A, Rubio B, Pallardo F, Catala MD. Rapid-rate transcranial magnetic stimulation of left dorsolateral prefrontal cortex in drug-resistant depression. Lancet. 1996 Jul 27;348(9022):233-7. doi: 10.1016/s0140-6736(96)01219-6. PMID 8684201
- [Background] Chung SW, Hill AT, Rogasch NC, Hoy KE, Fitzgerald PB. Use of theta-burst stimulation in changing excitability of motor cortex: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2016 Apr;63:43-64. doi: 10.1016/j.neubiorev.2016.01.008. Epub 2016 Feb 3. PMID 26850210
- [Background] Jelic MB, Milanovic SD, Filipovic SR. Differential effects of facilitatory and inhibitory theta burst stimulation of the primary motor cortex on motor learning. Clin Neurophysiol. 2015 May;126(5):1016-23. doi: 10.1016/j.clinph.2014.09.003. Epub 2014 Sep 16. PMID 25281475
- [Background] Chung SW, Hoy KE, Fitzgerald PB. Theta-burst stimulation: a new form of TMS treatment for depression? Depress Anxiety. 2015 Mar;32(3):182-92. doi: 10.1002/da.22335. Epub 2014 Nov 28. PMID 25450537
- [Background] Plewnia C, Pasqualetti P, Grosse S, Schlipf S, Wasserka B, Zwissler B, Fallgatter A. Treatment of major depression with bilateral theta burst stimulation: a randomized controlled pilot trial. J Affect Disord. 2014 Mar;156:219-23. doi: 10.1016/j.jad.2013.12.025. Epub 2013 Dec 28. PMID 24411682
- [Background] Prasser J, Schecklmann M, Poeppl TB, Frank E, Kreuzer PM, Hajak G, Rupprecht R, Landgrebe M, Langguth B. Bilateral prefrontal rTMS and theta burst TMS as an add-on treatment for depression: a randomized placebo controlled trial. World J Biol Psychiatry. 2015 Jan;16(1):57-65. doi: 10.3109/15622975.2014.964768. Epub 2014 Nov 28. PMID 25430687
- [Background] Daskalakis ZJ. Theta-burst transcranial magnetic stimulation in depression: when less may be more. Brain. 2014 Jul;137(Pt 7):1860-2. doi: 10.1093/brain/awu123. Epub 2014 May 15. No abstract available. PMID 24833712
- [Background] Thut G, Pascual-Leone A. A review of combined TMS-EEG studies to characterize lasting effects of repetitive TMS and assess their usefulness in cognitive and clinical neuroscience. Brain Topogr. 2010 Jan;22(4):219-32. doi: 10.1007/s10548-009-0115-4. Epub 2009 Oct 28. PMID 19862614
- [Background] Holtzheimer PE 3rd, McDonald WM, Mufti M, Kelley ME, Quinn S, Corso G, Epstein CM. Accelerated repetitive transcranial magnetic stimulation for treatment-resistant depression. Depress Anxiety. 2010 Oct;27(10):960-3. doi: 10.1002/da.20731. PMID 20734360
- [Background] Fung PK, Robinson PA. Neural field theory of synaptic metaplasticity with applications to theta burst stimulation. J Theor Biol. 2014 Jan 7;340:164-76. doi: 10.1016/j.jtbi.2013.09.021. Epub 2013 Sep 21. PMID 24060620
- [Background] Biswal B, Yetkin FZ, Haughton VM, Hyde JS. Functional connectivity in the motor cortex of resting human brain using echo-planar MRI. Magn Reson Med. 1995 Oct;34(4):537-41. doi: 10.1002/mrm.1910340409. PMID 8524021
- [Background] Greicius MD, Krasnow B, Reiss AL, Menon V. Functional connectivity in the resting brain: a network analysis of the default mode hypothesis. Proc Natl Acad Sci U S A. 2003 Jan 7;100(1):253-8. doi: 10.1073/pnas.0135058100. Epub 2002 Dec 27. PMID 12506194
- [Background] Fox MD, Snyder AZ, Vincent JL, Corbetta M, Van Essen DC, Raichle ME. The human brain is intrinsically organized into dynamic, anticorrelated functional networks. Proc Natl Acad Sci U S A. 2005 Jul 5;102(27):9673-8. doi: 10.1073/pnas.0504136102. Epub 2005 Jun 23. PMID 15976020
- [Background] Greicius MD, Supekar K, Menon V, Dougherty RF. Resting-state functional connectivity reflects structural connectivity in the default mode network. Cereb Cortex. 2009 Jan;19(1):72-8. doi: 10.1093/cercor/bhn059. Epub 2008 Apr 9. PMID 18403396